CLINICAL TRIAL: NCT04267081
Title: Two-stage, Two-arm, Open-Label Phase II Study of Venetoclax in Combination With Azacytidine in Acute Myeloid Leukemia Patients Selected Using Ex Vivo Drug Sensitivity Screening
Brief Title: Study of Venetoclax in Combination With Azacytidine in AML Patients Selected Using Ex Vivo Drug Sensitivity Screening
Acronym: VenEx
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Mika Kontro, Principal Investigator, Helsinki University Central Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FLG-V001
Record Dates: First submitted 2020-02-07; First posted 2020-02-12 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML; Venetoclax; Azacytidine; Drug Sensitivity Screening
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax

STUDY DESIGN:
Intervention Model Description: This is a multicenter two-stage, two-arm, open label phase II study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (de novo AML) (Experimental): This arm will recruit the patients with de novo AML unfit for conventional chemotherapy. In validation cohort all the participants will receive azacytidine-venetoclax. In study cohort the patients with ex vivo resistance to venetoclax will be excluded from the study therapy.
  All patients in validation and study cohorts (ARM1 and ARM2) will receive azacytidine and venetoclax. The purpose for the validation cohort is to validate the specificity and sensitivity of the ex vivo drug testing. Patients exhibiting ex vivo sensitivity and receiving azacytidine-venetoclax in validation cohort are analyzed also for study cohort.
  Interventions: Drug: Venetoclax
- Arm 2 (relapsed, refractory or secondary AML) (Experimental): This arm will recruit the patients with relapsed, refractory or secondary AML. In validation cohort all the participants will receive azacytidine-venetoclax. In study cohort the patients with ex vivo resistance to venetoclax will be excluded from the study therapy.
  All patients in validation and study cohorts (ARM1 and ARM2) will receive azacytidine and venetoclax. The purpose for the validation cohort is to validate the specificity and sensitivity of the ex vivo drug testing. Patients exhibiting ex vivo sensitivity and receiving azacytidine-venetoclax in validation cohort are analyzed also for study cohort.
  Interventions: Drug: Venetoclax

INTERVENTIONS:
Drug: Venetoclax — Ex vivo venetoclax sensitivity testing is used for patient selection.
  Other Names: Ex vivo drug sensitivity testing

SUMMARY:
This is a multi center two-stage, two-arm, open label phase II study of venetoclax in combination with azacytidine in acute myeloid leukemia patients selected for therapy with ex vivo venetoclax sensitivity screening. This study will characterize the usability of ex vivo drug sensitivity testing for patient selection for selecting the responsive patients for venetoclax therapy. The exploratory study will aim to find novel combinations for overcoming resistance as well as finding/validating biomarkers for both sensitivity and resistance.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Patients who present with one of the following (except acute promyelocytic leukemia):

   * De novo or secondary AML patients who are non-fit for standard induction therapy (see below)
   * Relapsed or refractory AML patients following at least 1 line of prior therapies (see below)
3. Ex vivo sensitivity testing performed to assess venetoclax sensitivity

   1. Validation cohort: All participants are treated with venetoclax+azacitidine irrespective of the ex vivo screening results.
   2. Study cohort: Only the participants exhibiting ex vivo sensitivity to venetoclax are included to study therapy.
4. Participant must have ECOG Performance status ≤ 2 for participants ≥ 75 years of age OR ≤ 3 for participants ≥ 18 to 74 years of age
5. Leukocyte count < 25 x10E9/l. Hydroxyurea use is permitted to meet this criterion.
6. Participant must have adequate renal function as demonstrated by a calculated creatinine clearance ≥ 30 mL/min; determined by the Cockcroft Gault formula.
7. Participant must have adequate liver function as demonstrated by

   1. alanine aminotransferase (ALT) ≤ 4.0 × ULN
   2. bilirubin ≤ 1.5 × ULN
8. Specific inclusion criteria for participants non-fit for standard chemotherapy

   Participant must be:

   ≥ 70 years of age OR ≥ 18 to 69 years of age and ineligible for intensive chemotherapy meeting at least one of the criteria following:
   * Clinically significant comorbidities, reflected at least 1 of:

     * Left ventricular ejection fraction (LVEF) < 50%.
     * Lung diffusion capacity for carbon monoxide (DLCO) ≤ 65% of expected.
     * Forced expiratory volume in 1 second (FEV1) ≤ 65% of expected.
     * Chronic stable angina or congestive heart failure controlled with medication.
     * Alanine aminotransferase (ALT) 3.0-4.0 × ULN
   * Other contraindication(s) to anthracycline therapy (must be documented)
   * Adverse risk karyotype associated with poor outcome with standard chemotherapy
   * Patient's refusal from intensive chemotherapy
9. Specific inclusion criteria for relapsed patients

   Participant must be ≥ 55 years of age with non-CBF AML relapse OR ≥ 18 of age and meeting at least one of the criteria following:
   * Not candidate for intensive chemotherapy (see the criteria 8.)
   * The duration of remission < 12 months.
   * Relapse after allogeneic transplantation.
   * 2nd (or higher) relapse.
10. Specific inclusion criteria for refractory patients The patients who fail to achieve a complete or partial remission after induction chemotherapy (two cycles of chemotherapy containing cytarabine or clofarabine, in compilation with topoisomerase II inhibitor (e.g. anthracycline or mitoxantrone)

Exclusion Criteria:

1. Participant has acute promyelocytic leukemia (APL)
2. The leukemic cell content (blast percentage) in bone marrow/peripheral blood (depending which is used for drug sensitivity testing) is ≤ 10 %
3. ECOG >3 (see also inclusion criteria 4)
4. Participant has known CNS involvement with AML (note: CSF or radiological investigations are not required without clinical suspicion)
5. Participant with known HIV infection or active hepatitis B virus (HBV), or hepatitis C virus (HCV) infection that is not controlled with anti-viral medication.
6. Participant has cardiovascular disability status of New York Heart Association Class ≥ 2. Class 2 is defined as cardiac disease in which participants are comfortable at rest but ordinary physical activity results in palpitations, fatigue, dyspnea, or anginal pain.
7. Evidence of clinically significant condition(s) that in the opinion of the investigator would adversely affect his/her participation in this study (including but not limited to):

   1. Participant has a chronic respiratory disease that requires continuous oxygen use
   2. Systemic uncontrolled infection requiring therapy (viral, bacterial or fungal)
   3. Malabsorption syndrome or other condition that precludes enteral route of administration.
   4. Uncontrolled GVHD.
8. Participant has a history of other malignancies prior to study entry, with the exception of previous malignancy treated with curative intent.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2020-02-12 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Complete remission (CR)/complete remission rate with incomplete hematologic recovery (CRi) rate in study cohort after three cycles. | The bone marrow is examined at the end of Cycle 3. Each cycle is 28 days.

SECONDARY OUTCOMES:
The correlation of ex vivo venetoclax sensitivity and specific responses: Overall Survival (OS), Duration of Response (DOR), Event-free Survival (EFS) and Minimal Residual Disease (MRD) status. | Through study completion, an average of 3 years
The correlation of venetoclax blood concentrations to specific responses: Overall Survival (OS), Duration of Response (DOR), Event-free Survival (EFS) and Minimal Residual Disease (MRD) status. | Through study completion, an average of 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- HelsinkiUCH, Helsinki, Uusimaa, Finland

REFERENCES:
- [Derived] Kytola S, Vanttinen I, Ruokoranta T, Partanen A, Holopainen A, Saad J, Kuusisto MEL, Koskela S, Raty R, Itala-Remes M, Vastrik I, Suvela M, Parsons A, Porkka K, Wennerberg K, Heckman CA, Jalkanen T, Huttunen T, Ettala P, Rimpilainen J, Siitonen T, Pyorala M, Kuusanmaki H, Kontro M. Ex vivo venetoclax sensitivity predicts clinical response in acute myeloid leukemia in the prospective VenEx trial. Blood. 2025 Jan 23;145(4):409-421. doi: 10.1182/blood.2024024968. PMID 39357056
- [Derived] Kuusanmaki H, Kytola S, Vanttinen I, Ruokoranta T, Ranta A, Huuhtanen J, Suvela M, Parsons A, Holopainen A, Partanen A, Kuusisto MEL, Koskela S, Raty R, Itala-Remes M, Vastrik I, Dufva O, Siitonen S, Porkka K, Wennerberg K, Heckman CA, Ettala P, Pyorala M, Rimpilainen J, Siitonen T, Kontro M. Ex vivo venetoclax sensitivity testing predicts treatment response in acute myeloid leukemia. Haematologica. 2023 Jul 1;108(7):1768-1781. doi: 10.3324/haematol.2022.281692. PMID 36519325